CLINICAL TRIAL: NCT00696124
Title: Phase 1, Dose-Escalation Study to Assess the Safety and Tolerability of VM202 (Engensis) in Subjects With Critical Limb Ischemia
Brief Title: Safety Study of Gene Therapy in Treating Critical Leg Ischemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Helixmith Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: US 06-1-001
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Results first posted 2024-10-18 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-08

CONDITIONS: Critical Limb Ischemia
Keywords: lower leg ischemia; peripheral artery disease
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (Experimental): 2 mg dose VM202. The first half of the total dose given on Day 1 and the second half on Day 15.
  Interventions: Biological: VM202 2 mg
- Cohort 2 (Experimental): 4 mg dose VM202. The first half of the total dose given on Day 1 and the second half on Day 15.
  Interventions: Biological: VM202 4 mg
- Cohort 3 (Experimental): 8 mg dose VM202. The first half of the total dose given on Day 1 and the second half on Day 15.
  Interventions: Biological: VM202 8 mg
- Cohort 4 (Experimental): 16 mg dose VM202. The first half of the total dose given on Day 1 and the second half on Day 15.
  Interventions: Biological: VM202 16 mg

INTERVENTIONS:
Biological: VM202 2 mg — 2 mg intramuscular injection with the first half of the total dose given on Day 1 and the second half on Day 15
  Arms: Cohort 1
Biological: VM202 4 mg — 4 mg intramuscular injection, with half of the total dose given on Day 1 and the second half given on Day 15
  Arms: Cohort 2
Biological: VM202 8 mg — 8 mg intramuscular injection. The first half of the total dose given on Day 1 and the second half on Day 15.
  Arms: Cohort 3
Biological: VM202 16 mg — 16 mg dose intramuscular injection. The first half of the total dose given on Day 1 and the second half on Day 15.
  Arms: Cohort 4

SUMMARY:
The purpose of this study is to determine the safety, tolerability and preliminary efficacy of intramuscular injections of VM202 for subjects with critical limb ischemia.

Subjects selected for this study will have critical limb ischemia that has not responded to standard therapy with symptoms including pain at rest and/or ischemic ulcers.

DETAILED DESCRIPTION:
The study will consist of four (4) cohorts with a total of 3 subjects enrolled in each cohort to VM202.For each dose cohort, VM202 will be administered as a local intramuscular injection in 2 divided doses with a 2-week interval between the injections. Preliminary efficacy (hemodynamic assessments), safety and tolerability will be evaluated at Baseline (screening) and at designated time points throughout the study.

After the first subject in each cohort completed Day 30 (±2 days), and before the Day 15 dosing of the other 2 subjects in the same cohort, an interim safety evaluation was performed with the submission of safety data to the Data Safety Monitoring Committee.

All four dose cohorts will be followed for up to 5 years from the time of the first dose of study drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between 20 and 90 years of age
* Have critical limb ischemia (Rutherford Class 4 and 5) and considered not a candidate for bypass graft surgery or percutaneous angioplasty due to co-morbid conditions, failure of previous surgical or interventional procedures or caliber of grafting arteries. Critical Limb ischemia is defined as

  1. Stable symptoms on standard therapy including anti-platelet agents, vascular rheologic agents, cilostazol, anticoagulant and pain medication for 30 days.
  2. Pain at rest and/or ischemic ulcers for a minimum of 4 weeks.
* Have diagnostic angiography of the affected limb in the last 12 months demonstrating a significant occlusion of one more of the following arteries: iliac, superficial femoral, popliteal, and one or more infra-popliteal arteries.
* Have a resting ankle systolic pressure (in either the dorsalis pedis or posterior tibial arteries) of less than or equal to 60mmHg or a resting toe systolic pressure of less than or equal to 40 mmHg in the affected limb.
* Be willing to maintain current drug therapy for peripheral arterial disease throughout the course of the study including anti-platelet and statin inhibitor treatment
* Be capable of understanding and complying with the protocol and signing the informed consent document prior to being subjected to any study related procedures
* Women who are surgically sterile or at least 1 year postmenopausal or who have been practicing adequate contraception for at least 12 weeks prior to entering the study. If the subject is of child-bearing potential, she must have a negative serum pregnancy test result prior to study enrollment and must agree to repeat pregnancy screening tests during the study
* If the subject or the subject's partner(s) is of child bearing potential, the subject and the subject's partner(s) must agree to use a "double barrier" method of birth control while participating in this study.

Exclusion Criteria:

* Subjects who have undergone a revascularization procedure or sympathectomy within 12 weeks prior to study entry that remains patent. A failed revascularization procedure in the previous 4 weeks is acceptable.
* Subjects with grade 3 (hemorrhages, exudates) or grade 4 (papilledema) retinopathy.
* Subjects currently receiving immunosuppressive medications, chemotherapy, radiation therapy.
* Subject with aorta-iliac occlusion (greater than 75%).
* Subjects that will require amputation within 4 weeks of randomization.
* Subjects with any co-morbid conditions likely to interfere with assessment of safety or efficacy or with an estimated life expectancy of less than 6 months
* Subjects with history of drug (defined as illicit drug use) or a history of alcohol abuse (defined as regular or daily consumption of more than 4 alcoholic drinks per day) within the past 3 months.
* Subjects with a current history or new screening finding of malignant neoplasm except for basal cell carcinoma of the skin and squamous cell carcinoma of the skin (if excised and no evidence of recurrence).
* Subjects with evidence of active infection (e.g. cellulitis, osteomyelitis) or deep ulceration exposing bone or tendon in the extremity planned for treatment.
* Subjects with a clinically significant abnormality in routine hematology, urinalysis, chemistry, liver function or other laboratory tests, including HIV, Hepatitis B, Cytomegalovirus, hepatitis C virus, Venereal Disease Research Laboratory test, prostate-specific antigen, and chorio-embryonic antigen, or signs of malignant neoplasm by radiological imaging tests, including chest radiography at Screening or Day 1. Specific laboratory exclusion criteria include the following:

  1. Hemoglobin less than 9.0 g/dL
  2. White Blood Cell count less than 3,000 cells/mm3
  3. Platelet count less than 75,000 platelets/uL
  4. Fasting glucose greater than 250 mg/dL
  5. AST and/or ALT greater than 3X upper limit of normal
* Subjects with any other condition that in the opinion of the investigator might put the subject at risk or interfere with his/her participation.
* Subjects unwilling or unable to comply with the protocol or to cooperate fully with the investigator or site personnel.
* Subjects that have received any other investigational drug within the 30 days prior to study drug administration or will receive such a drug during the time frame of this study.
* Subjects with uncontrolled hypertension defined as systolic blood pressure greater than 200 mmHg or diastolic blood pressure greater than 115 mmHg at Baseline evaluation.
* Subjects with advanced liver disease including decompensated cirrhosis, jaundice, ascites, or bleeding varices.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-04-03 (Actual); Primary Completion 2009-10-19 (Actual); Study Completion 2023-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Henry, MD, Principal Investigator — Minneapolis Heart Institute Foundation
Locations (1):
- Minneapolis Heart Institute Foundation/ Abbott Northwestern Hospital, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Henry TD, Hirsch AT, Goldman J, Wang YL, Lips DL, McMillan WD, Duval S, Biggs TA, Keo HH. Safety of a non-viral plasmid-encoding dual isoforms of hepatocyte growth factor in critical limb ischemia patients: a phase I study. Gene Ther. 2011 Aug;18(8):788-94. doi: 10.1038/gt.2011.21. Epub 2011 Mar 24. PMID 21430785
- See also: non-viral plasmid-encoding HGF in critical limb ischemia — https://www.nature.com/articles/gt201121

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Engensis 2 mg (VM202). The 2 mg intramuscular injection was given on Day 1 (first half of the total dose) and Day 15 (the second half of the total dose)
- Cohort 2: Engensis 4 mg (VM202). The 4 mg intramuscular injection was given on Day 1 (first half of the total dose) and Day 15 (the second half of the total dose)
- Cohort 3: Engensis 8 mg (VM202). The 8 mg intramuscular injection was given on Day 1 (first half of the total dose) and Day 15 (the second half of the total dose)
- Cohort 4: Engensis 16 mg (VM202). The 16 mg intramuscular injection was given on Day 1 (first half of the total dose) and Day 15 (the second half of the total dose)
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (15.1) | 70.0 (5.3) | 70.3 (9.0) | 63.7 (20.8) | 67.8 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 2 | 5
  Male | 2 | 2 | 2 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 2 | 3 | 3 | 3 | 11
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Treatment-Emergent Adverse Events.
Description: Treatment-emergent adverse events defined as adverse events after the first dose of Engensis (Day 1) through Day 365
Time Frame: Day 1 to Day 365
Population: Safety population included all subjects who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 3 | 3 | 3 | 3
Participants
  Subjects with at least one TEAE | 3 | 3 | 3 | 3
  Infections and Infestations | 2 | 1 | 3 | 1
  Urinary tract infection | 2 | 0 | 1 | 1
  Upper respiratory infection | 0 | 1 | 1 | 0
  Cellulitis | 1 | 0 | 0 | 0
  Chronic sinusitis | 0 | 1 | 0 | 0
  Wound infection | 0 | 0 | 1 | 0
  General Disorders and Administration Site Conditions | 2 | 0 | 1 | 0
  Chest pain | 1 | 0 | 0 | 0
  Injection site bruising | 1 | 0 | 0 | 0
  Pyrexia | 0 | 0 | 1 | 0
  Musculoskeletal and Connective Tissue Disorders | 0 | 1 | 1 | 1
  Pain in extremity | 0 | 1 | 1 | 0
  Muscle spasms | 0 | 0 | 0 | 1
  Musculoskeletal pain | 0 | 0 | 0 | 1
  Neoplasms Benign, Malignant and Unspecified (Including Cysts and Polyps) | 1 | 1 | 1 | 0
  Biliary adenoma | 0 | 1 | 0 | 0
  Colon cancer | 0 | 0 | 1 | 0
  Metastases to liver | 1 | 0 | 0 | 0
  Small cell lung cancer stage unspecified | 1 | 0 | 0 | 0
  Respiratory, Thoracic and Mediastinal Disorders | 1 | 2 | 0 | 0
  Rhonchi | 1 | 0 | 0 | 0
  Throat irritation | 0 | 1 | 0 | 0
  Wheezing | 0 | 1 | 0 | 0
  Vascular Disorders | 1 | 0 | 2 | 0
  Peripheral arterial occlusive disease | 0 | 0 | 2 | 0
  Haematoma | 1 | 0 | 0 | 0
  Hypotension | 0 | 0 | 1 | 0
  Blood and Lymphatic System Disorders | 0 | 1 | 1 | 0
  Anaemia | 0 | 1 | 1 | 0
  Cardiac Disorders | 1 | 1 | 0 | 0
  Bundle branch block left | 1 | 0 | 0 | 0
  Cyanosis | 0 | 1 | 0 | 0
  Gastrointestinal Disorders | 1 | 0 | 1 | 0
  Gastric ulcer | 0 | 0 | 1 | 0
  Ileus | 1 | 0 | 0 | 0
  Investigations | 1 | 0 | 1 | 0
  Blood creatinine increased | 0 | 0 | 1 | 0
  Blood glucose increased | 0 | 0 | 1 | 0
  Glucose urine present | 0 | 0 | 1 | 0
  International normalized ratio increased | 0 | 0 | 1 | 0
  Prostatic specific antigen increased | 1 | 0 | 0 | 0
  Skin and Subcutaneous Tissue Disorders | 0 | 1 | 0 | 1
  Erythema | 0 | 1 | 0 | 0
  Pruritus | 0 | 0 | 0 | 1
  Skin ulcer | 0 | 0 | 0 | 1
  Injury, Poisoning and Procedural Complications | 1 | 0 | 0 | 0
  Tongue injury | 1 | 0 | 0 | 0
  Psychiatric Disorders | 1 | 0 | 0 | 0
  Confusional state | 1 | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline in Pain Visual Analog Scale
Description: Pain intensity was assessed by subjects marking a place on a 100 mm Visual Analog Scale ranging from 0 = no pain to 100 = worst possible pain. The distance from 0 to the mark was to be measured in millimeters (0 to 100 mm).
Time Frame: Days 15, 28, 59, 91, 180, and 365
Population: The Intent-to-Treat population included all subjects who received at least one dose of study drug medication and had at least one post-dose assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 3 | 3 | 3 | 3
score on a scale
  Baseline (Day 0) Actual values only | 66.7 (20.79) | 64.3 (12.90) | 38.3 (45.79) | 50.3 (20.31)
  Day 15 | -0.3 (19.30) | -20.7 (22.19) | 1.7 (9.87) | 7.0 (19.67)
  Day 28 | 4.0 (14.42) | -53.7 (18.88) | 8.7 (7.23) | -15.3 (3.06)
  Day 59 | -8.3 (30.01) | -52.0 (10.39) | 13.0 (9.00) | -26.3 (14.57)
  Day 91 | -3.3 (29.02) | -56.3 (9.07) | 1.0 (11.36) | 0.0 (38.11)
  Day 180 | -12.3 (22.68) | -63.3 (12.22) | 31.0 (55.15) | -29.7 (19.55)
  Day 365 | -13.7 (35.5) | -63.3 (13.61) | 37.5 (58.69) | 4.3 (9.87)

3. Secondary Outcome: Change From Baseline in Ankle Brachial Index
Description: The Ankle Brachial Index is the ratio of the systolic blood pressure at the ankle to the systolic blood pressure in the upper arm (brachial). Outcome measure is the Change in Baseline from Day 0 (Baseline) to Actual visit Days (Days 15, 28, 59, 91, 180 and 365).
Time Frame: Days 15, 28, 59, 91, 180, and 365
Population: Intent-to-treat population, defined as all subjects who received at least one dose of study drug and had at least one post-dose assessment
Measure: Mean (Standard Deviation); unit: Ratio Systolic BP-Change ankle to arm
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 3 | 3 | 3 | 3
Ratio Systolic BP-Change ankle to arm
  Baseline (Day 0) Actual values only | 0.35 (0.10) | 0.35 (0.04) | 0.44 (0.06) | 0.57 (0.43)
  Day 15 | 0.10 (0.12) | 0.05 (0.04) | 0.02 (0.02) | 0.04 (0.14)
  Day 28 | 0.0 (0.14) | 0.14 (0.07) | -0.06 (0.17) | -0.08 (0.38)
  Day 59 | 0.08 (0.08) | 0.14 (0.14) | -0.10 (0.17) | 0.13 (0.24)
  Day 91: number analyzed (Participants) | 3 | 2 | 3 | 2
  Day 91 | 0.14 (0.09) | 0.05 (0.13) | -0.03 (0.03) | 0.09 (0.32)
  Day 180: number analyzed (Participants) | 3 | 3 | 2 | 3
  Day 180 | 0.06 (0.14) | 0.07 (0.11) | -0.05 (0.08) | 0.15 (0.05)
  Day 365: number analyzed (Participants) | 3 | 3 | 1 | 3
  Day 365 | 0.12 (0.06) | 0.21 (0.15) | 0.13 (NA) — No SD available for 1 participant | 0.13 (0.19)

4. Secondary Outcome: Change From Baseline in Toe Brachial Index
Description: Toe brachial index is the ratio of the systolic blood pressure of the toes to the systolic blood pressure in the upper arm (brachial). Outcome measure is the Change in Ratio for Baseline from Day 0 (Baseline) to Actual visit Days (Days 15, 28, 59, 91, 180 and 365).
Time Frame: Baseline and Days 1,15,28,59,91,180,and 365
Population: Intent-to-treat population defined as all subjects who received at least one dose of study drug and had at least one post-dose assessment
Measure: Mean (Standard Deviation); unit: Ratio Systolic BP-Change toe to arm
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 3 | 3 | 3 | 3
Ratio Systolic BP-Change toe to arm
  Baseline (Day 0) Actual values only | 0.16 (0.04) | 0.19 (0.01) | 0.18 (0.11) | 0.22 (0.26)
  Day 15 | 0.0 (0.07) | 0.07 (0.05) | -0.05 (0.13) | 0.22 (0.01)
  Day 28 | -0.01 (0.09) | -0.01 (0.02) | -0.02 (0.08) | 0.03 (0.01)
  Day 59 | 0.08 (0.09) | 0.05 (0.05) | -0.04 (0.09) | 0.14 (0.03)
  Day 91: number analyzed (Participants) | 3 | 2 | 3 | 2
  Day 91 | 0.04 (0.15) | 0.06 (0.04) | -0.08 (0.08) | 0.12 (0.06)
  Day 180: number analyzed (Participants) | 3 | 3 | 2 | 3
  Day 180 | 0.05 (0.06) | 0.10 (0.12) | 0.01 (0.12) | 0.01 (0.22)
  Day 365: number analyzed (Participants) | 3 | 3 | 1 | 3
  Day 365 | 0.10 (0.07) | 0.14 (0.11) | -0.08 | 0.11 (0.03)

5. Secondary Outcome: Change From Baseline in Transcutaneous Oxygen Pressure
Description: At Screening, transcutaneous oxygen pressure was measured at pre-defined locations on the anterior and posterior calf and dorsum of the foot. The limb/chest Transcutaneous Oxygen Pressure index was calculated by using the lower of the distal limb measurements
Time Frame: Days 1 to 365
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 3 | 3 | 3 | 3
mmHg
  Baseline (Day 0) Actual values only | 48.7 (12.10) | 47.0 (18.03) | 38.3 (11.02) | 70.7 (4.51)
  Day 91 | 10.0 (8.72) | 4.3 (13.87) | 2.7 (13.32) | -1.3 (5.13)
  Day 180 | 15.0 (10.54) | 13.0 (6.24) | 10.0 (11.31) | -16.3 (21.96)
  Day 365 | 9.0 (7.81) | 7.3 (7.64) | 25.5 (2.12) | -3.7 (7.37)

ADVERSE EVENTS:
Time Frame: Day 1 through Day 365
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 3/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=3) | Cohort 4 (N=3)
Metastases to Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small Cell Lung Cancer - Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biliary Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=3) | Cohort 4 (N=3)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 1 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Bundle Branch Block Left (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cyanosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glucose urine present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostatic specific antigen increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Chronic Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2009-09-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT00696124/Prot_000.pdf
  • Statistical Analysis Plan (2008-01-10): https://cdn.clinicaltrials.gov/large-docs/24/NCT00696124/SAP_001.pdf